CLINICAL TRIAL: NCT05754632
Title: The Impact of Blood Flow Restriction Training in Adolescents After ACL Reconstruction: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-139
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Injuries; Knee Injuries; Quadriceps Muscle Atrophy
Keywords: physical therapy; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Intervention Model Description: A single randomized control trial will compare the use of exercises augmented with BFRT with quantitative measurements of strength and patient-reported outcomes. A total of 40 youth and adolescent patients undergoing a surgical procedure for ACLR and subsequent physical therapy at our institution will be recruited for this study.
  Patients will be randomized into one of two groups using computer randomization for allocation: the intervention group receiving BFRT as part of physical therapy, and the control group will follow the institution's standard ACLR rehabilitation protocol. Both groups will follow a time- and criterion-based standardized rehabilitation protocol. The primary outcomes will be isometric and isokinetic knee peak torque and limb symmetry indices. Secondary outcomes will be quadriceps hypertrophy via mid-thigh circumference and patient-reported outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BFR Intervention Group (Experimental): In addition to the standard ACL rehabilitation protocol, the experimental group will complete 2 exercises using the Delfi BFR cuff 2x/week for 8 weeks during their treatment session at Connecticut Children's Sports Physical Therapy on the second post-operative visit. Cuff size will be determined by patient thigh circumference Limb occlusion pressure will be determined in supine position and all exercises will be completed at 80% occlusion.
  Long Arc Quadriceps (LAQ) progression Shuttle progression Post-op visit 2- 2 weeks Quadriceps Set Standing Straight Leg Raise 2 weeks-4 weeks Available range LAQ Standing terminal knee extension 4 weeks-8 weeks LAQ (0-90°) Single Limb Shuttle/Leg Press
  Interventions: Device: Blood Flow Restriction using Delfi Personalized Tourniquet System
- No Intervention/Control Group (No Intervention): In addition to the standard ACL rehabilitation protocol, the control group will complete the same exercises as the experimental group starting on the second post-operative visit.
  Long Arc Quadriceps (LAQ) progression Shuttle progression Post-op visit 2- 2 weeks Quadriceps Set Standing Straight Leg Raise 2 weeks-4 weeks Available range LAQ Standing terminal knee extension 4 weeks-8 weeks LAQ (0-90°) Single Limb Shuttle/Leg Press

INTERVENTIONS:
Device: Blood Flow Restriction using Delfi Personalized Tourniquet System — The Delfi Tourniquet System is designed to be used in conjunction with exercise. The system automatically determines the degree of occlusion and allows for safe regulation of pressure. Patients will then complete exercises with the use of this device.
  Other Names: FDA Establishment Registration Number 9681444. Device Listing Number E127474. Classification Number 878.5910. Product Code KCY. 510(k) Exempt. MID: XCDELMED1099VAN
  Arms: BFR Intervention Group

SUMMARY:
While there are a number studies that have reported on the use of blood flow restriction training (BFRT) in the adult population, there is limited information about the use of BFRT in the adolescent population. This study aims to evaluate the use of BFRT in conjunction with traditional anterior ligament reconstruction (ACLR) rehabilitation in adolescents.

The purpose of this study is to compare the addition of a BFRT based exercise protocol to a standard ACL rehabilitation protocol in adolescents. Does the addition of BFRT-based exercise improve strength, hypertrophy, and patient reported outcomes after ACLR in the adolescent population?

DETAILED DESCRIPTION:
A single randomized control trial will compare the use of exercises augmented with BFRT with quantitative measurements of strength and patient-reported outcomes. A total of 40 youth and adolescent patients undergoing a surgical procedure for ACLR and subsequent physical therapy at our institution will be recruited for this study. Patients will be randomized into one of two groups using computer randomization for allocation: the intervention group receiving BFRT as part of physical therapy, and the control group will follow the institution's standard ACLR rehabilitation protocol. Both groups will follow a time- and criterion-based standardized rehabilitation protocol. The primary outcomes will be isometric and isokinetic knee peak torque and limb symmetry indices. Secondary outcomes will be quadriceps hypertrophy via mid-thigh circumference and patient-reported outcomes.

Target Population Adolescent patients between the ages of 12 and 18 will be recruited at the time of surgery, specifically, those that participate in sports who are undergoing primary ACLR reconstruction at Connecticut Children's

Study Group and Control Group Inclusion Criteria

· Prior to surgery participated in > 50 hours/year of level I or II sports as defined by Noyes et al and planned to return to prior level.

Level I Sports (4-7 days/week) Jumping, hard pivoting, cutting (basketball, volleyball, football, soccer, gymnastics, skiing. wrestling) Running, twisting, turning (racquet sports, baseball, hockey) Level II sports (1-3 days/week) Jumping, hard pivoting, cutting (basketball, volleyball, football, soccer, gymnastics, skiing. wrestling) Running, twisting, turning (racquet sports, baseball, hockey)

* Completion of postoperative rehabilitation following standard protocols
* Orthopedic surgical intervention and physical therapy completed at Connecticut Children's.

ELIGIBILITY:
Inclusion Criteria:

* Prior to surgery participated in >50 hours/year of level I or II sports as defined by Noyes et al and planned to return to prior level.

Level I Sports (4-7 days/week) Jumping, hard pivoting, cutting (basketball, volleyball,football, soccer, gymnastics, skiing. wrestling)

* Level II sports (1-3 days/week) Jumping, hard pivoting, cutting (basketball, volleyball,football, soccer, gymnastics, skiing. wrestling)
* Completion of postoperative rehabilitation following standard protocols
* Orthopedic surgical intervention and physical therapy completed at Connecticut Children's.

Exclusion Criteria:

* An additional lower extremity injury at time of knee injury or previous surgical intervention on the knee (ipsilateral and contralateral)
* Multiple ligament ruptures or trauma
* Weight bearing restrictions for greater than 4 weeks after surgery due to concomitant pathology such as meniscal root/radial repair, chondral pathology, or multi-ligament pathology
* Follow-up surgical procedures including, but not limited to, post-operative arthrofibrosis Inability to attend regular physical therapy sessions (≥80% of patient treatment sessions and all assessment visits
* Contraindications to performing BFRT including known history of central or peripheral neurologic impairments, cardiac or metabolic condition or history of deep vein thrombosis (DVT).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | Change in range of motion at Pre-op, 3 months post-op, 6 months post-op, 9 months post-op
  Active knee range of motion: Knee AROM will be measured in supine position using a goniometer and standardized procedures reported by Norkin and White
Isometric Quad strength Peak Torque | Change in strength at Pre-op, 3 months post-op, 6 months post-op, 9 months post-op
  Isometric strength testing to measure peak torque quadriceps strength (unit: ft-lbs) as reported by isokinetic dynamometer on involved and uninvolved limb.
Isometric Quadriceps Strength limb symmetry index | Change in strength at Pre-op, 3 months post-op, 6 months post-op, 9 months post-op
  Quadriceps limb symmetry index is calculated by taking the values from outcome 1. [ ( peak torque quadriceps involved limb (ft/lbs)/ peak torque quadriceps uninvolved limb (ft-lbs))*100] as reported by isokinetic dynamometer. This value is expressed as a percentage. 100% would equal perfect symmetry.
Isometric Hamstring Strength Peak Torque | Change in strength at Pre-op, 3 months post-op, 6 months post-op, 9 months post-op
  Isometric strength testing to measure peak torque hamstring strength (unit: ft-lbs) as reported by isokinetic dynamometer on involved and uninvolved limb.
Isometric Hamstring Strength Limb Symmetry Index | Change in strength at Pre-op, 3 months post-op, 6 months post-op, 9 months post-op
  Hamstring limb symmetry index is calculated by taking the values from outcome 3 [ ( peak torque hamstring involved limb (ft/lbs) / peak torque hamstring uninvolved limb (ft-lbs))*100] as reported by isokinetic dynamometer. This value is expressed as a percentage.100% would equal perfect symmetry.
Isokinetic Quadriceps strength | Change in strength at 6 months and 9 months post-op
  Isokinetic strength testing to measure peak torque quadriceps strength (unit: ft-lbs) as reported by isokinetic dynamometer on involved and uninvolved limb.
Isokinetic Quadriceps Strength limb symmetry index | Change in strength at 6 months and 9 months post-op
  Quadriceps limb symmetry index is calculated by taking the values from outcome 1. [ ( peak torque quadriceps involved limb (ft/lbs)/ peak torque quadriceps uninvolved limb (ft-lbs))*100] as reported by isokinetic dynamometer. This value is expressed as a percentage. 100% would equal perfect symmetry.
Isokinetic Hamstrings Strength | Change in strength at 6 months and 9 months post-op
  Isokinetic strength testing to measure peak torque hamstring strength (unit: ft-lbs) as reported by isokinetic dynamometer on involved and uninvolved limb.
Isokinetic Hamstring Strength limb symmetry index | Change in strength at 6 months and 9 months post-op
  Hamstring limb symmetry index is calculated by taking the values from outcome 1. [ ( peak torque quadriceps involved limb (ft/lbs)/ peak torque quadriceps uninvolved limb (ft-lbs))*100] as reported by isokinetic dynamometer. This value is expressed as a percentage. 100% would equal perfect symmetry.

SECONDARY OUTCOMES:
Quadriceps Hypertrophy | Change in strength at Pre-op, 8 weeks, 3months post-op, 6months, 9 months post-op
  Thigh Circumference measured at location 10cm superior to patella and measured in cm comparing involved to uninvolved lower extremity
Pediatric International Knee Documentation Committee | Tracking change at Pre-op, 3months post-op, 6 months post-op, 9 months post-op. 2 years post-op
  Patient Reported Outcome Measure- Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Knee Outcomes and Osteoarthritis Scale | Tracking change at Pre-op, 3months post-op, 6 months post-op, 9 months post-op. 2 years post-op
  Patient Reported Outcome Measure- The score is a percentage score from 0 to 100, with 0 representing extreme problems and 100 representing no problems. This scoring direction, 100 indicating no problems
Anterior Cruciate Ligament- Return to Sport after Injury | Tracking change at Pre-op, 3months post-op, 6 months post-op, 9 months post-op. 2 years post-op
  Patient Reported Outcome Measure- The scores range from 0 to 100, with higher scores representing patients who are more ready to return to sport
Tegner Activity Scale | changes from pre-operative, 9 months, and 2 years post-operative
  Tegner activity scale will measure sport level- higher level equals higher sport competitive level

CONTACTS AND LOCATIONS:
Overall Officials: Adam Weaver, PT, DPT, Principal Investigator — Physical Therapist
Locations (1):
- Connecticut Children's Sports Physical Therapy, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT05754632/Prot_000.pdf